CLINICAL TRIAL: NCT02001519
Title: A Phase ll Trial of Impact of Additional 4 Cycles of Cisplatin (CDDP4) in Patients With Triple Negative Breast Cancer Not Achieving Clinical CR After 4 Cycles of Neoadjuvant Adriamycin Plus Cyclophosphamide
Brief Title: Additional 4 Cycles of Cisplatin (CDDP4) in Patients With Triple Negative Breast Cancer for Neoadjuvant Chemotherapy
Acronym: PACER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Bae Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNBC AC-CDDP
Record Dates: First submitted 2012-07-05; First posted 2013-12-05 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adriamycin,cytoxan, cisplatin (Experimental): 4 cycles of Adriamycin 60 mg/m2 and Cyclophosphamide 600 mg/m2 every 3 weeks followed by 4 cycles of cisplatin 75 mg/m2 every 3 weeks
  Interventions: Drug: AC4-CDDP4

INTERVENTIONS:
Drug: AC4-CDDP4 — 4 cycles of Adriamycin 60 mg/m2 and Cyclophosphamide 600 mg/m2 every 3 weeks 4 cycles of cisplatin 75 mg/m2 every 3 weeks

SUMMARY:
Achievement of pathologic complete response is important prognosticator to predict long term outcome in triple negative cancer. The efficacy of adding 4 cycles of cisplatin (CDDP4) is to be investigated whether addtional pathologic complete response is achieved for those triple negative breast cancer patients who recieved 4 cycles of adriamycin with cyclophosphamide(AC4) but did not reach clinical complete response during the course of neoadjuvant therapy.

DETAILED DESCRIPTION:
First outcome measures (analysis) :at the time of surgery,

Second outcome measures:

2019 August, 5 year Overall Survival, Disease free survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven breast cancer
2. Age, at least 20 years
3. ER/PR/HER2 (negative/negative/negative

   * ER/PR negative: nuclear reaction < 1%, Allred score 0 or 2
   * HER2 negative: HER2; IHC (immunohistochemistry) 0,1+ or FISH/SISH (-) in case of IHC 2+
4. Clinically stage II or III with histologically proven lymph-node involvement (T >1.5 cm or lymph node [LN] >1.5 cm)
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. No prior hormonal treatment, chemotherapy or radiotherapy is allowed.
7. Adequate hematologic, liver and kidney function
8. Written informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. Prior chemotherapy or radiotherapy for any malignancy
3. Stage T4d; inflammatory breast cancer
4. No primary tumor (T0)
5. Documented history of cardiac disease contraindicating anthracyclines
6. Currently active infection

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | up to 36 weeks
  Rate of pCR (as defined by NSABP [National Surgical Adjuvant Breast and Bowel Project] criteria - absence of invasive disease in the breast [ypT0]) at the time of surgery.

SECONDARY OUTCOMES:
Overall response rate (ORR) by radiologic evaluation | up to 36 weeks
  after completion of chemotherapy Overall objective clinical response rate = CR (complete response) + PR (partial response) rate, measured by US (or MRI) and assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Complete metabolic response (CMR) rate after 2 cycles of AC | up to 12 weeks
  after 2 cycles of AC
3 year disease free survival (3yr-DFS) | 3 years
Rate of breast conservation | up to 36 weeks
  after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea